CLINICAL TRIAL: NCT04924179
Title: A Phase II, Single-arm, Open-label, Single Center Study of Tislelizumab Combined With Fruquintinib and SBRT as A Third-line and Posterior Line Treatment in Patients With Advanced Colorectal Cancer
Brief Title: Tislelizumab Combined With Fruquintinib and SBRT as Athird-line and Posterior Line Treatment in Patients With Advanced CRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, Huazhong University of Science and Technology, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C113
Record Dates: First submitted 2021-06-03; First posted 2021-06-11 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Patients With Advanced Metastatic Colorectal Cancer
MeSH Terms: interventions — tislelizumab; HMPL-013; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab plus Fruquintinib and SBRT (Experimental)
  Interventions: Drug: Tislelizumab plus Fruquintinib and SBRT

INTERVENTIONS:
Drug: Tislelizumab plus Fruquintinib and SBRT — Fruquintinib:5mg ,qd,po, d1-d14, 21 days for a cycle;Tislelizumab Injection:200mg，IV,d1,21 days for a cycle;SBRT:8-10Gy×5F,qod,in 10 days.

SUMMARY:
A Phase II Study to Assess the Efficacy and Safety of Tislelizumab Combined With Fruquintinib and SBRT as A third-line and Posterior Line Treatment in Patients With Advanced Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written Informed Consent Form (ICF) prior to any study specific procedures
2. Age ≥ 18 years, ≤75 years
3. Histologically or cytologically confirmed advanced Stage IV primary colorectal cancer
4. One or more organs metastases, and the metastases are suitable for SBRT according to the evaluation of the researchers;
5. At least two or more standard systemic therapies prior treatment (based on Fu, oxaliplatin, irinotecan, bevacizumab and cetuximab) of cytotoxic chemotherapy, treatment failure or intolerable toxicities
6. ECOG 0-1
7. Patients must have measurable lesions
8. Expected overall survival ≥12 weeks
9. AST, ALT and alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN)，Serum bilirubin ≤ 1.5 x ULN，creatinine<ULN
10. Prothrombin time (PT), international standard ratio (INR) ≤1.5 × ULN
11. Patients are allowed to have received radiotherapy, but the time from entering the group must be more than 4 weeks, and the currently selected radiotherapy lesions and evaluable lesions must be lesions that have not received radiotherapy
12. Women of childbearing age must be willing to use adequate contraceptives during the study period of drug treatment

Exclusion Criteria:

1. Patients have received anti-PD-1 / PD-L1 immunotherapy or other immunoexperimental drugs
2. Patients with severe autoimmune diseases: active inflammatory bowel disease (including Crohn's disease and ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (such as Wegener's granuloma), etc
3. Risk factors of intestinal perforation: active diverticulitis, abdominal abscess, gastrointestinal obstruction, abdominal cancer or other known risk factors of intestinal perforation
4. Known hereditary or acquired bleeding (such as coagulation dysfunction) or thrombotic tendency, such as hemophilia patients
5. Aspirin (> 325 mg / day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel (≥ 75 mg) and cilostazol are currently used or have been used recently (within 10 days before the start of study treatment)
6. Thrombosis or embolism events such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction) and pulmonary embolism occurred within 6 months before the start of the study
7. The researchers believe that the patient has a lesion and needs emergency palliative radiotherapy / emergency surgery (spinal cord compression, brain hernia, pathological fracture)
8. Known active infection and active tuberculosis infection were not included in the group; However, patients with hepatitis B virus (HBV) and hepatitis C virus (HCV) infection can be included in the group if their condition is stable after antiviral treatment;
9. There is evidence of pneumoperitoneum that cannot be explained by puncture or recent surgery;
10. Patients with history of hepatic encephalopathy;
11. Participated in the clinical trials of other drugs that have not been approved or marketed in China and received the corresponding experimental drug treatment within 2 weeks before enrollment
12. systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg regardless of any antihypertensive drugs; Or patients need more than two antihypertensive drugs
13. Patients have untreated central nervous system metastasis
14. Received any operation or invasive treatment or operation (except venous catheterization, puncture and drainage, etc.) within 4 weeks before enrollment
15. Patients have not recovered from all toxicities associated with prior anti-tumor therapy ,to acceptable baseline status, or a National Cancer Institute Common Terminology Criteria for Adverse Events(NCI CTCAE v5.0) Grade of 0 or 1, except for alopecia and oxaliplatin induced neurotoxicity ≤ 2 , and the previous surgery did not recover completely
16. Dysphagia or known malabsorption of drugs
17. Active gastric and duodenal ulcer, ulcerative colitis or uncontrolled hemorrhage in GI
18. Have evidence or history of bleeding tendency within 2 months after enrollment, the researcher assessed that moderate or severe bleeding tendency was not suitable for enrollment
19. Patients had other malignant tumors in the past 5 years or at the same time (except for the cured skin basal cell carcinoma and cervical carcinoma in situ);
20. Pregnant or lactating women
21. Allergic to Surufatinib/Vinorelbine
22. History of immunodeficiency, including HIV positive, other acquired or congenital immunodeficiency diseases, or organ transplantation
23. Patients with acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before admission; Or a history of arterial thrombosis or deep venous thrombosis
24. There are concomitant diseases (such as severe hypertension, diabetes, thyroid disease, active infection, etc.) that seriously endanger the safety of patients or affect the completion of the study, or any laboratory abnormalities that are not suitable for participating in the clinical trial according to the judgment of the researcher
25. Active autoimmune disease or history of autoimmune disease with possible recurrence (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism);
26. Immunosuppressive agents or systemic hormones were used 14 days before the start of the study to achieve the purpose of immunosuppression (dose > 10mg / day prednisone or other therapeutic hormones)
27. Known to have a history of severe allergy to any monoclonal antibody or antiangiogenic target drug
28. Serious psychological or mental disorders that may affect the compliance study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 16 months
  To assess the efficacy of Tislelizumab Combined With Fruquintinib and SBRT for patients with advanced colorectal cancer by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 16 months
  CR + PR rate according to the RECIST version 1.1 guidelines.
Disease control rate (DCR) | up to 16 months
  Disease control rate (DCR):CR + PR + SD rate according to the RECIST version 1.1 guidelines.
Overall survival (OS) | up to 36 months
  The time interval between the start date of study drug and the date of death (any cause)
AEs | up to 36 months
  Adverse reactions refer to the occurrence and development of diseases in the process of using drugs according to normal usage and dosage to prevent, diagnose or treat diseases.Adverse reactions unrelated to the purpose of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No